CLINICAL TRIAL: NCT03268057
Title: Phase 1b/Study of VX15/2503 in Combination With Avelumab in Advanced Non-small Cell Lung Cancer
Brief Title: VX15/2503 in Combination With Avelumab in Advanced Non-small Cell Lung Cancer
Acronym: CLASSICAL-Lung
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vaccinex Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VX15/2503-04
Record Dates: First submitted 2017-08-11; First posted 2017-08-31 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-Small-Cell Lung; Carcinoma; Advanced; VX15/2503; Semaphorin 4D; SEMA4D; safety tolerability; pharmacokinetics; monoclonal antibody; IO Failure; Immunotherapy Failure; Decline Chemo
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma | interventions — avelumab

STUDY DESIGN:
Intervention Model Description: A dose escalation phase based on the use of a 3 + 3 design and treament of up to 6 subjects in each of three VX15/2503 dose levels; a fixed dose of avelumab will be employed. Once the recommended phase two dose is determined, subjects will receive that dose of VX15/205 combined with avelumab moving forward.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VX15/2503 + avelumab (Experimental): VX15/2503 at a concentration of 5 mg/kg, 10 mg/kg or 20 mg/kg with a fixed dose of avelumab at 10 mg/kg, administered intravenously on a bi-weekly dosing cycle.
  Interventions: Drug: VX15/2503 + avelumab

INTERVENTIONS:
Drug: VX15/2503 + avelumab — Dose escalation will begin at 5 mg/kg of VX15/2503 and will increase up to 20 mg/kg with a constant dose of avelumab at 10 mg/kg. A recommended phase II dose of VX15/2503 will be determined and then utilized in the expansion phase with 10 mg/kg of avelumab.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of IV administration of VX15/2503 in combination with a fixed dose of avelumab in patients with advanced non-small cell lung cancer. The dose escalation portion of the study will determine the maximum tolerated dose (MTD) of VX15/2503 administered in combination with avelumab.

DETAILED DESCRIPTION:
This is a phase 1b/2 study, designed to evaluate the safety, tolerability, and efficacy of VX15/2503 in combination with avelumab in subjects diagnosed with advanced (stage IIIB/IV) NSCLC who have either progressed on first or second-line systemic anticancer therapy or who have declined treatment with first or second-line system anticancer therapy. The primary objective (Dose Escalation Phase) is to evaluate the safety and tolerability of ascending doses of VX15/2503 Q2W in combination with avelumab 10mg/kg Q2W. The second primary objective (Dose Expansion Phase) is to evaluate safety and tolerability of the recommended phase 2 dose of VX15/2503 administered in combination with 10 mg/kg avelumab Q2W. The secondary objectives include (Dose Expansion Phase), a preliminary estimate of efficacy using the following in accordance with Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, Objective Response (OR), Duration of Response (DoR) and Progression-Free Survival (PFS), as well as making a preliminary estimate of efficacy using the following in accordance with iRECIST, OR, DoR and PFS. Additional secondary objectives are to characterize the pharmacokinetics profile of VX15/2503 and avelumab administered Q2W in combination, evaluate the immunogenicity of VX15/2503 and avelumab administered Q2W and evaluate VX15/2503 and avelumab pharmacodynamics markers including but not limited to receptor occupancy. Exploratory objectives include identification of candidate biomarkers of activity and biomarkers that may predict response to treatment with combination therapy of VX15/2503 and avelumab.

Enrollment will involve approximately 62 individuals who are 18 years of age or older with advanced non-small cell lung cancer. The study will be divided into two phases, dose escalation with up to 18 Immunotherapy naive subjects and dose expansion with up to 50 subjects (up to 22 subjects that are Immunotherapy naive and up to 28 subjects that have failed on Immunotherapy). Subjects that are enrolled in the dose escalation phase may continue into the dose expansion phase, as long as there is no evidence of disease progression. The subjects entering the dose expansion phase from dose escalation, may have their dose increased to the recommend phase 2 dose, once it is determined. Any subjects that have evidence of disease progression will be taken off of treatment and will have a post treatment safety follow-up visit 10 weeks after last treatment. Subjects that have discontinued study drug will also continue to be followed every 3 months for survival, or lost to follow-up. It is estimated that the study will take approximately 33 months between first subject enrolled and last subject visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. Signed informed consent prior to the performance of any study-specific procedures, including fresh tumor biopsies.
3. Histologically or cytologically proven advanced (stage IIIB/IV) NSCLC subjects. Subjects in the Dose Escalation Phase must be immunotherapy naïve.
4. i. Subjects in the Dose Escalation Phase must have either progressed on or declined standard first-line therapy. Subjects with fewer than 3 lines of prior palliative systemic anti-cancer therapy are eligible.

   ii. Subjects in the Dose Expansion Phase must have progressed on a minimum of 2 cycles of standard of care platinum-based chemotherapy with or without immunotherapy, standard of care immunotherapy without chemotherapy or must have declined standard of care first-line treatment options. Subjects with fewer than 3 lines of prior palliative systemic anti-cancer therapy are eligible.
5. Subjects previously treated with systemic adjuvant/neoadjuvant therapy, other than immunotherapy are also eligible for the Dose Escalation Phase. Subjects previously treated with standard of care systemic adjuvant/neoadjuvant therapy are also eligible for the Dose Expansion Phase.
6. Measureable disease as defined by the RECIST 1.1.
7. Availability of archival or fresh tumor specimen that is suitable for analysis. Acceptable samples must have been acquired using core needle biopsy or excisional biopsy. Samples that were acquired using fine needle aspiration are not acceptable.
8. Tumor lesion accessible for biopsy after the start of treatment. (Note: this lesion should be separate from measurable lesions that will be used for response assessment.)
9. ECOG performance status (PS) score 0-1.
10. Left ventricular ejection fraction > 50%
11. Tumors lack activating epidermal growth factor receptor (EGFR) mutations, ROS-1, or ALK rearrangement (no EGFR or ALK testing is required if a subject has a KRAS mutation or squamous cell histology)..
12. Has adequate bone marrow, renal and hepatic function based upon laboratory tests as follows:

    * Absolute neutrophil count > 1500/µL
    * Platelet count > 100 x 103/µL
    * Hemoglobin > 9 g/dL, transfusion permitted
    * Total bilirubin < 1.5 x upper limit of normal (ULN) (or < 3 x ULN for subjects with Gilbert's syndrome)
    * Creatinine clearance ≥ 50 mL/min on the basis of the Cockcroft-Gault glomerular filtration rate calculation
    * AST < 2.5 x ULN (5.0 x ULN in the presence of liver metastasis)
    * ALT < 2.5 x ULN (5.0 x ULN in the presence of liver metastasis).
13. Highly effective contraception (i.e., methods with a failure rate of less than 1 % per year) for both male and female subjects if the risk of conception exists (Note: The effects of the trial treatment on the developing human fetus are unknown; thus, women of childbearing potential and men must agree to use highly effective contraception, defined in Protocol Appendix 9.3, or as stipulated in national or local guidelines. Highly effective contraception must be used for the duration of trial treatment, and at least for 60 days after stopping trial treatment or 6 months after stopping chemotherapy [or per label]. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this trial, the treating physician should be informed immediately).

Exclusion Criteria:

1. Prior therapy with any antibody or drug targeting T-cell coregulatory proteins (immune checkpoints), such as PD-1, PD-L1, or cytotoxic T lymphocyte antigen-4 in the Dose Escalation Phase only.
2. Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on Investigator's judgment are acceptable.
3. Concurrent anticancer treatment within 28 days before the start of trial treatment (e.g., cytoreductive therapy, radiotherapy [with the exception of palliative bone directed radiotherapy]; immune therapy, or cytokine therapy, except for erythropoietin.
4. Major surgery within 28 days before the start of trial treatment (excluding prior diagnostic biopsy); or use of any investigational drug within 28 days before the start of trial treatment.
5. Subjects receiving immunosuppressive agents (such as steroids) for any reason should be tapered off these drugs before initiation of the trial treatment (with the exception of subjects with adrenal insufficiency, who may continue corticosteroids at physiologic replacement dose, equivalent to ≤ 10 mg prednisone daily). Note: Previous or ongoing administration of systemic steroids for the management of an acute allergic phenomenon is acceptable as long as it is anticipated that the administration of steroids will be completed in 14 days, or that the daily dose after 14 days will be ≤10 mg per day of prednisone or equivalent.
6. Previous malignant disease other than the target malignancy to be investigated in this trial within the last 5 years (with the exception of adequately treated non-melanoma skin cancers, carcinoma in situ of skin, bladder, cervix, colon/rectum, breast, or prostate) unless a complete remission without further recurrence was achieved at least 2 years prior to study entry and the subject was deemed to have been cured with no additional therapy required or anticipated to be required.
7. Rapidly progressive disease disease (i.e. disease progression before or at the time of first tumor assessment, 8 - 12 weeks after initiation of systemic anti-cancer therapy).
8. ECOG performance status score ≥ 2.
9. Women who are pregnant or breastfeeding.
10. History of pneumonitis or other interstitial lung disease
11. Active or history of any autoimmune disease including colitis and inflammatory bowel disease (subjects with diabetes Type I, vitiligo, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible) or immunodeficiencies.
12. Vaccination within 4 weeks of the first dose of avelumab and while on study is prohibited except for administration of inactivated vaccines (e.g. inactivated influenza vaccines).
13. Significant acute or chronic infection including, among others: Known history of human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome. Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection (defined as, HBV surface antigen positive and HBV core antibody positive with reflex to positive HBV DNA or HBV core antibody positive alone with reflex to positive HBV DNA or positive HCV antibody with reflex to positive HCV RNA).
14. Central nervous system malignancy, the known presence of untreated or symptomatic CNS metastases. Subjects with treated brain metastasis must be stable and off steroids and anti-convulsants for at least 1 month prior to the start of study treatment. Subjects with suspected brain metastases at Screening should have a CT/MRI of the brain prior to study entry.
15. A history of hypersensitivity to other humanized monoclonal antibodies.
16. Significant cardiovascular disease (New York Heart Association Class II or greater), myocardial infarction within the 6 months prior to study entry, unstable angina, or cerebral vascular accident / stroke (< 6 months prior to enrollment), or serious uncontrolled cardiac arrhythmia requiring medication / active intervention, corrected QT interval [QTc] prolongation of >= 470ms and/or prior diagnosis of congenital long QT syndrome.
17. Legal incapacity or limited legal capacity.
18. Current alcohol or drug abuse.
19. Any psychiatric condition that would prohibit the understanding or rendering of informed consent.
20. Prior organ transplantation or allogeneic bone marrow transplantation.
21. Any uncontrolled medical condition (for example, inflammatory bowel disease, uncontrolled asthma), which, in the opinion of the Investigator, might impair the subject's tolerance of trial treatment or confound interpretation of study assessments.
22. Inability to comply with visit schedule or other protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Dose Escalation Phase: Number of subjects with dose-limiting toxicities (DLT)s at each dose level | 21 Days for Each Escalation Phase
  DLTs will be described and graded according to the Common Terminology Criteria Adverse Events version 4.03 (CTCAE v4.03) and according to the specific MedRA terms from immune mediated AEs
Dose Expansion Phase: Frequency and type of adverse events (AE)s | 2 Years
  Safety assessments will be performed on a regular basis using physical examination, spontaneous AE reporting, scheduled and unscheduled laboratory assessments, and other diagnostic evaluations as indicated. Adverse events will be reported using the Common Terminology Criteria Adverse Events version 4.03 (CTCAE v4.03).

SECONDARY OUTCOMES:
Dose Expansion Phase: Objective Response (OR) | 2 Years
  This is defined as complete response (CR) or partial response (PR) according to RECIST 1.1 from first dose until documented confirmed disease progression.
Dose Expansion Phase: Duration of Response (DoR) | 2 Years
  This is defined, for subjects with an objective response, as the time from first confirmed documented objective response (CR or PR) to the date of first confirmed documented objective progression of disease (PD) or death.
Dose Expansion Phase: Progression Free Survival (PFS) | 2 Years
  This is defined as the time from first dose to the date of the first confirmed documented objective progression of disease (PD) or death
Dose Expansion Phase: Peak serum concentration (Cmax) of VX15/2503 and avelumab | 2 Years
  PK Parameter
Dose Expansion Phase: Area under the serum concentration versus time curve (AUC) of VX15/2503 and avelumab | 2 Years
  PK Parameter
Dose Expansion Phase: Half-life of VX15/2503 and avelumab | 2 Years
  PK Parameter
Dose Expansion Phase: Immunogenicity of VX15/2503 and avelumab as measured by frequency and titer of human anti human antibodies | 2 Years
  Anti Drug Antibodies (ADA)
Dose Expansion Phase: Receptor occupancy of VX15/2503 and avelumab as measured by a flow cytometry based saturation assay | 2 Years
  PD Parameter
Dose Expansion Phase: Cellular SEMA4D levels as measured by flow cytometry | 2 Years
  PD Parameter
Dose Expansion Phase: Total soluble SEMA4D levels as measured by ELISA | 2 Years
  PD Parameter

CONTACTS AND LOCATIONS:
Overall Officials: John E Leonard, PhD, Study Director — Vaccinex Inc.
Locations (11):
- United States (11):
  - Highlands Oncology Group, PA, Fayetteville, Arkansas
  - University of California Los Angeles (UCLA), Los Angeles, California
  - Mayo Clinic, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Northwell Health Cancer Institute, Lake Success, New York
  - University of Rochester, Rochester, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Virginia Cancer Specialists, PC, Fairfax, Virginia

REFERENCES:
- [Background] Patnaik A, Weiss GJ, Leonard JE, Rasco DW, Sachdev JC, Fisher TL, Winter LA, Reilly C, Parker RB, Mutz D, Blaydorn L, Tolcher AW, Zauderer M, Ramanathan RK. Safety, Pharmacokinetics, and Pharmacodynamics of a Humanized Anti-Semaphorin 4D Antibody, in a First-In-Human Study of Patients with Advanced Solid Tumors. Clin Cancer Res. 2016 Feb 15;22(4):827-36. doi: 10.1158/1078-0432.CCR-15-0431. Epub 2015 Oct 7. PMID 26446947
- [Background] Evans EE, Jonason AS Jr, Bussler H, Torno S, Veeraraghavan J, Reilly C, Doherty MA, Seils J, Winter LA, Mallow C, Kirk R, Howell A, Giralico S, Scrivens M, Klimatcheva K, Fisher TL, Bowers WJ, Paris M, Smith ES, Zauderer M. Antibody Blockade of Semaphorin 4D Promotes Immune Infiltration into Tumor and Enhances Response to Other Immunomodulatory Therapies. Cancer Immunol Res. 2015 Jun;3(6):689-701. doi: 10.1158/2326-6066.CIR-14-0171. Epub 2015 Jan 22. PMID 25614511
- [Background] Seymour L, Bogaerts J, Perrone A, Ford R, Schwartz LH, Mandrekar S, Lin NU, Litiere S, Dancey J, Chen A, Hodi FS, Therasse P, Hoekstra OS, Shankar LK, Wolchok JD, Ballinger M, Caramella C, de Vries EGE; RECIST working group. iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics. Lancet Oncol. 2017 Mar;18(3):e143-e152. doi: 10.1016/S1470-2045(17)30074-8. Epub 2017 Mar 2. PMID 28271869
- [Derived] Shafique MR, Fisher TL, Evans EE, Leonard JE, Pastore DRE, Mallow CL, Smith E, Mishra V, Schroder A, Chin KM, Beck JT, Baumgart MA, Govindan R, Gabrail NY, Spira AI, Seetharamu N, Lou Y, Mansfield AS, Sanborn RE, Goldman JW, Zauderer M. A Phase Ib/II Study of Pepinemab in Combination with Avelumab in Advanced Non-Small Cell Lung Cancer. Clin Cancer Res. 2021 Jul 1;27(13):3630-3640. doi: 10.1158/1078-0432.CCR-20-4792. Epub 2021 Apr 5. PMID 33820783
- See also: Safety, Pharmacokinetics, and Pharmacodynamics of a Humanized Anti-Semaphorin 4D Antibody, in a First-In-Human Study of Patients with Advanced Solid Tumors. — https://www.ncbi.nlm.nih.gov/pubmed/26446947
- See also: Antibody Blockade of Semaphorin 4D Promotes Immune Infiltration into Tumor and Enhances Response to Other Immunomodulatory Therapies — https://www.ncbi.nlm.nih.gov/pubmed/?term=Antibody+Blockade+of+Semaphorin+4D+Promotes+Immune+Infiltration+into+Tumor+and+Enhances+Response+to+Other+Immunomodulatory+Therapies